CLINICAL TRIAL: NCT03582423
Title: The Efficacy and Safety of Acupuncture for Alleviating Chemotherapy-induced Peripheral Neuropathy in Colorectal Cancer Patients: a Pilot Single-blinded, Randomized Sham-controlled Trial
Brief Title: Acupuncture for Chemotherapy-induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Zhong Lidan, Research Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKBU-YCH
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized, sham-acupuncture controlled trial
Who Masked: Participant
Masking Description: Subjects of both groups will be randomly assigned to receive either electro-acupuncture or control (sham) treatment. For randomization, simple, complete non-sequential random numbers will be generated in advance by a computer program in a block of four, and kept by the principal investigator. After a patient's eligibility is confirmed, a randomization number which corresponds to the group allocation will be provided to the acupuncturist by the PI. This arrangement will ensure that the clinical assessor and participants are blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electro-acupuncture group (Experimental): Eight acupoints are chosen: he gu (LI4), nei guan(PC6), qu chi (LI12), ba xie (EX-UE9), zu san li (ST36), san yin jiao (SP6), tai chung (LV3) and ba feng (EX-LE10). The use of ba xie (EX-UE9) and ba feng (EX-LE10) will be optional if skin lesions of hands and feet occurs due to Capecitabine (Xeloda).Disposable acupuncture needles will be inserted at a depth of 10-25mm into the points. We will deliver electrical stimulation with continuous waves at 2 Hz, at an intensity of each patient's minimum sensation of stimulation through the electrical acupuncture stimulation instrument to the points. The needles will be retained in position for 25 minutes.
  Interventions: Other: electro-acupuncture
- sham-acupuncture group (Placebo Comparator): Streitberger's non-invasive acupuncture needles (Gauge 8 × 1.2"/ 0.30 × 30mm) will be applied to serve as a sham control at the same acupoints with the same stimulation modality, except that the needles are only adhered to the skin by a small plastic ring instead of being inserted and the stimulation will be a "pseudo-stimulation"
  Interventions: Other: electro-acupuncture

INTERVENTIONS:
Other: electro-acupuncture — Eight acupoints are chosen: he gu (LI4), nei guan (PC6), qu chi (LI12), ba xie (EX-UE9), zu san li (ST36), san yin jiao (SP6), tai chung (LV3) and ba feng (EX-LE10). The use of ba xie (EX-UE9) and ba feng (EX-LE10) will be optional if skin lesions of hands and feet occurs due to Capecitabine (Xeloda).Disposable acupuncture needles will be inserted at a depth of 10-25mm into the points. We will deliver electrical stimulation with continuous waves at 2 Hz, at an intensity of each patient's minimum sensation of stimulation through the electrical acupuncture stimulation instrument to the points. The needles will be retained in position for 25 minutes.

SUMMARY:
In this study, a 24-week, single blinded, randomized controlled clinical trial will be conducted to examine the efficacy and safety of acupuncture for Chemotherapy Induced Peripheral Neuropathy (CIPN) in colorectal cancer patients in Hong Kong.

DETAILED DESCRIPTION:
This is a pilot single-blind, randomized, sham-controlled trial. 84 colorectal cancer patients will be randomly assigned to acupuncture group or control group. The duration of the treatment will be 12 weeks with 1 session per week and the follow-up period will be 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years old
* newly diagnosed with stage Ⅱto Ⅲcolorectal cancer
* who plan to receive 8 cycles of adjuvant oxaliplatin-based chemotherapy
* who have not received any acupuncture
* life expectancy of ≥ six months.

Exclusion Criteria:

* uncooperative subjects
* not be able to comprehend and communicate
* non-Chinese reading people
* having peripheral neuropathy caused by other diseases, for example, diabetes, stroke
* heart disease, for example, arrhythmia, heart failure, myocardial infarction or patients with pacemakers
* having a bleeding tendency
* be pregnant or lactating women
* having impaired hepatic or renal function
* using any pharmaceutical agents (for example, gabapentin, pregabalin), nutraceutical agents (for example, vitamin B6, vitamin E) and herbal medication for CIPN treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in scores of Functional Assessment of Cancer Therapy/Gynecology Oncology Group/Neurotoxicity (FACT/GOC-Ntx) questionnaire | 0,1,2,3,4,5,6,7,8,9,10,11,12,15,18,21,24 weeks
  FACT/GOC-Ntx includes 11 questions covering sensory neuropathy, motor neuropathy, hearing neuropathy, and dysfunction associated with neuropathy. It results in a cumulative score ranging from 0 to 44, with the higher scores reflecting worse neuropathy symptoms. It will be assessed every week during 12-week treatment and the post-trial access will be performed at 15th, 18th, 21st and 24th week.

SECONDARY OUTCOMES:
Changes in scores of numerical rating scale (NRS) of numbness/pain score in hands and feet | 0,1,2,3,4,5,6,7,8,9,10,11,12,15,18,21,24 weeks
  patients will be asked to rate their average neuropathy symptoms within one week, on an 0 to 10 scale (0 = no symptoms; 10 = worst possible symptoms), those <4 of 10 NRS will be considered as mild CIPN while ≥4 of 10 NRS will be considered as moderate to severe CIPN. It will be assessed every week during 12-week treatment and the post-trial access will be performed at 15th, 18th, 21st and 24th week.
Changes in scores of European Organization for Research and Treatment of Cancer (EORCTC) Quality of Life Questionnaire (QLQ-C30) | 0,3,6,9,12,15,18,21,24 weeks
  It is a 30-items questionnaire assessing five functional scales (physical, role, cognitive, emotional and social), three symptoms scales (fatigue, pain, nausea and vomiting), and other symptoms and problem in cancer patients (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties).It will be assessed every 3 weeks during 12-week treatment and the post-trial access will be performed at 15th, 18th, 21st and 24th week.
Changes in scores of Body Constitution of Chinese Medicine | 0,12,24 weeks
  Constitution of Chinese Medicine Questionnaire has 60 items measuring the 9 body constitution types: gentleness, Qi-deficiency, Yang-deficiency, Yin-deficiency, phlegm-wetness, wetness- heat, blood-stasis, Qi-depression, and special diathesis. It will be assessed at the end of treatment (12th week) and at the end of follow-up (24th week).
Changes in response of vibration sense test | 0,1,2,3,4,5,6,7,8,9,10,11,12,15,18,21,24 weeks
  It is assessed by using the graduated Rydel-Seiffer tuning fork. It will be assessed every week during 12-week treatment and the post-trial access will be performed at 15th, 18th, 21st and 24th week.
Changes in response of light touch test | 0,1,2,3,4,5,6,7,8,9,10,11,12,15,18,21,24 weeks
  It is assessed with standard 10g monofilaments, contained within the Neuropen. It will be assessed every week during 12-week treatment and the post-trial access will be performed at 15th, 18th, 21st and 24th week.
Adverse events after treatment and follow up | 0,1,2,3,4,5,6,7,8,9,10,11,12,15,18,21,24 weeks
  Adverse events after treatment will be recorded and compared among the two groups. It will be assessed every week during 12-week treatment and the post-trial access will be performed at 15th, 18th, 21st and 24th week.

CONTACTS AND LOCATIONS:
Overall Officials: Bacon Ng, Ph.D, Study Director — Department of Chinese Medicine, Hospital Authority
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chan K, Lui L, Lam Y, Yu K, Lau K, Lai M, Lau W, Tai L, Mak C, Bian Z, Zhong LL. Efficacy and safety of electroacupuncture for oxaliplatin-induced peripheral neuropathy in colorectal cancer patients: a single-blinded, randomized, sham-controlled trial. Acupunct Med. 2023 Oct;41(5):268-283. doi: 10.1177/09645284221125421. Epub 2022 Nov 3. PMID 36325677
- [Derived] Chan K, Lui L, Yu K, Lau K, Lai M, Lau W, Ng B, Zhong LLD, Bian ZX. The efficacy and safety of electro-acupuncture for alleviating chemotherapy-induced peripheral neuropathy in patients with coloreactal cancer: study protocol for a single-blinded, randomized sham-controlled trial. Trials. 2020 Jan 9;21(1):58. doi: 10.1186/s13063-019-3972-5. PMID 31918748